CLINICAL TRIAL: NCT00595582
Title: Early Intervention in Mild Cognitive Impairment (MCI) With Curcumin + Bioperine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: For various reasons.
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, James C. Patterson, II, MD. Ph, Professor, Louisiana State University Health Sciences Center Shreveport
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LSU#H05-168; LSU#H05-168 (Other: LSU Health Sciences Center IRB)
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Other): Curcumin + Bioperine
  Interventions: Dietary Supplement: curcumin + bioperine

INTERVENTIONS:
Dietary Supplement: curcumin + bioperine — Subjects who are currently in the primary Mild Cognitive Impairment study will be asked to be treated with 5.4 grams of curcumin + bioperine per day (900 mg pills, two pills 3x/day with meals) for 24 months concordant with the last two years of the primary longitudinal Mild Cognitive Impairment study.
  Other Names: Life Extension Super Bio-Curcumin

SUMMARY:
This is an additional study to the primary Mild Cognitive Impairment (MCI) study (LSU#H04-049; NCT00243451)that is underway of PET detection of Mild Cognitive Impairment. This study has preliminary data that indicates objective analysis of PET brain image metabolic data is a sensitive marker for AD. The goal of this proposal is to determine the efficacy of curcumin in the treatment of MCI or mild Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
The specific aims of this study include:

* Determine if curcumin has an effect on neuropsychological scores in patients with MCI. Working Hypothesis: Patients with MCI that have evidence of objective memory impairment will have improvement on neuropsychological test scores.
* Determine if curcumin impacts the metabolic lesions found in patients who have MCI or may develop MCI. Working hypothesis: The metabolic lesions present that are consistent with the development of early AD will improve with curcumin treatment.

Patients diagnosed with MCI, patients who have metabolic lesions consistent with premorbid MCI, or mild AD and are currently enrolled in the primary MCI study (LSU#H04-049; NCT00243451) will be invited to participate in this clinical trial.

These subjects will be treated with 5.4 grams of curcumin per day (900 mg pills, two pills 3X/day with meals) with the inclusion of bioperine additive (formulated with the curcumin capsules) to improve bioavailability of the curcumin. Patients will be treated with curcumin/bioperine for 24 months concordant with the last two years of the three year longitudinal primary MCI study. Clinical endpoints will be change in neuropsychological scores, and size of metabolic lesions on the PET scan. Both of these measures will be recorded as part of the primary MCI study.

ELIGIBILITY:
MCI Inclusion Criteria:

MCI criteria met:

* Memory complaint
* Objective memory impairment based on test scores
* Normal general cognitive function.
* Intact Activities of Daily Living.
* Not demented.
* At least 10 years of education, or GED, or equivalent.
* Patients with ApoE4 positive homozygous or heterozygous status and/or first-degree relative with probable AD are preferred
* Age: 55-85
* Have normal or clinically unimportant physical exam,
* Able to give informed consent, or assent
* MRI findings must be normal or unremarkable for the age of the patient.

Exclusion Criteria:

* Other neuropsychiatric diagnoses
* Major medical illness including potential secondary causes of cognitive decline.
* Disease, combination of disease, or presentation that, in the clinician's judgment, could introduce intolerable variance into the PET brain scan image
* Current substance or alcohol dependence or history of same, and no alcohol or substance abuse within the last eight weeks.

Mild Alzheimer's Disease (AD) Inclusion criteria (patients):

* You must have a Mini Mental State Examination score of greater than 20.
* You must have one or more of these signs and symptoms of mild AD all of which impair function and are worsening over time:

  1. Cognitive impairment manifested as memory problems
  2. problems with language
  3. difficulty carrying out motor activities
  4. difficulty naming things
  5. problems planning or organizing
* You must have at least 10 years of education, or a GED, or its equivalent.
* Positive for the ApoE4 genetic marker through blood test, or meet all other inclusion/exclusion criteria without exception.
* Age: 55-85.
* Normal or clinically unimportant physical exam
* Able to give informed consent/assent
* If you take medications that have an effect on the brain, they will be closely monitored. You will be PET-scanned only after a 24-hour washout of this medication(s), but this medication(s) will be restarted immediately after the scan.

Mild Alzheimer's Disease (AD) Exclusion Criteria:

* Any problems related to the brain or mental disorders other than mild AD.
* You will get an MRI of your brain taken on the second visit, and a radiologist will read it. If there are any abnormal findings, you will be told, and these findings will be forwarded to your medical doctor. These findings may or may not result in your exclusion from the study.
* Any major medical illness
* Any disease, combination of disease, or presentation that, in the clinician's judgment, could introduce intolerable variance into the PET brain scan image.
* Current diagnosis of substance or alcohol dependence or a history of same and no alcohol or substance abuse within the last eight weeks.

MCI Inclusion criteria (controls)

* Normal cognitive screening exam.
* Age: 55-85.
* At least 10 years of education or GED, or equivalent.
* Socioeconomic status, age, and sex matched.
* Able to give informed consent, or assent
* Centrally acting medications will be closely tracked, patients on any such medications will be PET-scanned only after a 24-hour washout, with meds restarted immediately after the scan.

MCI Exclusion criteria (controls)

* First-degree relative with dementia or clinically relevant memory problems.
* Other Neuropsychiatric diagnoses
* Major medical illness
* Current or history of substance or alcohol dependence; no alcohol or substance abuse within the last eight weeks.
* MRI findings must be normal or unremarkable for the age of the patient.
* Disease, combination of disease, or presentation that, in the clinician's judgment, could introduce intolerable variance into the PET brain scan image

Dropout criteria (all):

* Adverse events intolerable to the patient that prevent continued involvement in the study.
* New onset medical disorder of such significance as to prohibit further involvement.
* Initiation or recurrence of alcohol or substance abuse/dependence.
* Subject withdraws consent for any reason.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Patterson, MD, PhD, Principal Investigator — LSU Health Sciences Center
Locations (1):
- Louisiana State University Health Sciences Center, Shreveport, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were initially recruited for an MCI study which was IRB approved 9-29-03 and subjects were recruited from a medical clinic and advertising.
Period: Overall Study
Arm/Group | Curcumin + Bioperine
Started | 10
Completed | 0
Not Completed | 10
Not completed — Pilot study that PI terminated | 2
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 2
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Curcumin + Bioperine
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 77.6 (5.83476)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7.0
  Male | 3.0
Region of Enrollment [Number; unit: participants]
  United States | 10.0

OUTCOME MEASURES:

1. Primary Outcome: Neuropsychological Scores in Patients With MCI or Mild AD.
Time Frame: within the next three years
Population: No data were collected as this study was terminated.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Curcumin + Bioperine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Curcumin + Bioperine
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Curcumin + Bioperine (N=10)
dyspepsia (Gastrointestinal disorders) | 2

LIMITATIONS AND CAVEATS:
2 patients withdrew due to Dyspepsia (intolerance to supplement).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes